CLINICAL TRIAL: NCT01802216
Title: Kidney and Periodontal Disease Study
Acronym: KAPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A119016
Record Dates: First submitted 2013-02-15; First posted 2013-03-01 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Chronic Kidney Disease; Periodontal Disease
Keywords: chronic kidney disease progression; periodontal disease; intensive periodontal disease treatment
MeSH Terms: conditions — Renal Insufficiency, Chronic; Periodontal Diseases | interventions — Tooth Exfoliation; Root Planing; Minocycline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control/Delayed Treatment (No Intervention): Baseline panoramic x-ray (Panorex) and complete oral examinations at every visit. Rescue scaling and root planing only to sites of periodontal disease progression (since prior examination) of greater than 3mm. Subjects will be informed of their assignment to the delayed treatment group and provided referral list of local dentists should patient not feel comfortable waiting until end of study for full intensive periodontal disease treatment. Written and verbal instruction in oral hygiene. Provision of oral hygiene supplies.
- Intensive periodontal disease treatment (Active Comparator): Baseline panoramic x-ray (Panorex) and complete oral examinations at every visit. Intensive periodontal disease treatment to include administration of local anesthetic to up to two quadrants for scaling and root planing with ultrasonic and hand instruments. Minocycline will be applied to any sites with probing depth >=5mm. Hopeless teeth in scaled quadrants will be extracted. Written and verbal instruction in oral hygiene. Provision of oral hygiene supplies.
  Interventions: Procedure: Scaling and root planing; Drug: Minocycline

INTERVENTIONS:
Procedure: Scaling and root planing — non-surgical periodontal disease treatment
  Other Names: Deep cleaning; Subgingival cleaning
  Arms: Intensive periodontal disease treatment
Drug: Minocycline — antibiotic microspheres
  Other Names: Arestin
  Arms: Intensive periodontal disease treatment

SUMMARY:
The purpose of this study is (1) to determine whether a 12-month trial of patients from underserved communities with clinically significant gum disease and kidney disease randomly assigned to intensive gum disease treatment or delayed treatment is feasible and (2) to determine the variability of various tests of kidney function and inflammation in response to intensive gum disease treatment.

DETAILED DESCRIPTION:
This is a randomized controlled pilot trial to two intention-to-treat treatment arms: intensive periodontal therapy or control-delayed periodontal therapy. The investigators' goals are to test the feasibility of conducting this trial among an underserved (mostly poor and low literacy) population and to determine the variability of renal and inflammatory biomarkers in response to intensive periodontal therapy over a 12 month period among participants with both chronic kidney disease (CKD) and significant periodontal disease.

Randomization will be restricted with respect to diabetes (a strong risk factor for causing/aggravating both CKD and periodontal disease) to prevent an imbalance between the two arms. The investigators will recruit 51 patients from the San Francisco General Hospital (SFGH) Renal Clinic. Participants will be assigned 2:1 to the intervention group for the intensive periodontal treatment protocol (n=34) or to the control/delayed treatment group for rescue periodontal treatment only with intensive treatment at the end of the study (n=17).

Hypothesis:

A large scale randomized controlled trial of intensive periodontal treatment among the underserved will be feasible (with respect to enrollment, randomization, adherence and variability in clinical outcomes).

Specific Aims:

1. To assess the feasibility of recruiting patients to this pilot trial.
2. To determine the variability of kidney biomarkers in response to periodontal disease treatment.

Statistical Analysis:

The investigators will calculate descriptive statistics (mean, standard deviation) of each clinical outcome which will include a traditional marker of kidney function (serum creatinine), markers of kidney structure [as glomerular injury (albuminuria) and tubular injury (neutrophil gelatinase-associated lipocalin (NGAL))]; a marker of vascular endothelial injury (asymmetrical dimethylarginine (ADMA)); and markers of systemic inflammation (IL-6 and C-reactive protein) measured at baseline, study month 4, and study month 12. The investigators will use repeated-measures generalized estimating equations (GEE) to compare changes in clinical outcomes over time within each treatment group and to compare differences between treatment groups taking individual change over time into account.

Sample Size Calculation:

This is a pilot study. To the investigators' knowledge, there are no existing data of the anticipated effect size of periodontal treatment to inform sample size calculations. However, because a primary aim is to determine the variability of various renal and inflammatory biomarkers, the investigators seek to enroll at least 30 subjects in the intervention arm of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-75 years
2. Speaks English or Spanish
3. At least two measurements of estimated glomerular filtration (eGFR) rate 15-59 ml/min/1.73m2 within the preceding 12 months
4. No eGFR increase by >= 50% in the preceding 6 months
5. Moderate/severe periodontal disease in accordance with the Centers for Disease Control and Prevention/American Academy of Periodontology definition

Exclusion Criteria:

General Exclusion Criteria. Subjects must NOT be:

1. Under age 20 or over age 75
2. Unable to understand and provide informed consent
3. Receiving current immunosuppressant therapy.
4. Receiving current anticoagulation therapy resulting in an elevated prothrombin time or an International Normalized Ratio (INR) greater than 2.0
5. Pregnant.

Oral Exclusion Criteria. Subjects must NOT:

1. Have fewer than 6 natural teeth
2. Requires antibiotic prophylaxis for dental procedures as defined by the 2007 American Heart Association guidelines (patients with prosthetic heart valves, those with prosthetic material used for cardiac valve repair, those who have had a history of infective endocarditis, or those with congenital heart defects repaired with prosthetic material).
3. Have severe dental disease defined as deep dental caries, endodontic involvement of one or more teeth, presence of abscesses of periodontal or endodontic origin, or dental conditions requiring immediate treatment.
4. Have any hard or soft tissue lesion requiring further evaluation and/or treatment.
5. Have known allergy to minocycline, tetracyclines, or polyglycolide polymers.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-02; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Grubbs, MD, MPH, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grubbs V, Garcia F, Vittinghoff E, Jue BL, Ryder M, Lovett DH, Offenbacher S, Taylor G, Ganz P, Bibbins-Domingo K, Powe NR. Nonsurgical Periodontal Therapy in CKD: Findings of the Kidney and Periodontal Disease (KAPD) Pilot Randomized Controlled Trial. Kidney Med. 2019 Dec 2;2(1):49-58. doi: 10.1016/j.xkme.2019.09.005. eCollection 2020 Jan-Feb. PMID 32734226

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled English and Spanish-speaking patients 20-75 years old receiving primary care within the San Francisco Community Health Network. Patients with chronic kidney disease, not on dialysis, and moderate to severe periodontal disease are invited to participate.
Pre-assignment Details: Participants are assigned in a 2:1 ratio to control or intensive treatment group, randomization is stratified by presence of diabetes. Enrollment began February 2014 until September 2016. 101 participants attended the in-person oral exam screening. 55 were randomized, 46 were excluded (41 did not meet periodontal disease criteria and 5 declined.
Period: Baseline
Arm/Group | Control/Delayed Treatment | Intensive Periodontal Disease Treatment
Started | 17 | 34
Completed | 17 | 34
Not Completed | 0 | 0
Period: 4 Month Visit
Arm/Group | Control/Delayed Treatment | Intensive Periodontal Disease Treatment
Started | 17 | 34
Completed | 14 | 30
Not Completed | 3 | 4
Not completed — Participant did not show to visit | 3 | 4
Period: 8 Month Visit
Arm/Group | Control/Delayed Treatment | Intensive Periodontal Disease Treatment
Started | 17 | 34
Completed | 14 | 29
Not Completed | 3 | 5
Not completed — Participant did not show to visit | 3 | 5
Period: 12 Month Visit
Arm/Group | Control/Delayed Treatment | Intensive Periodontal Disease Treatment
Started | 17 | 34
Completed | 14 | 30
Not Completed | 3 | 4
Not completed — Participant did not show to visit | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control/Delayed Treatment | Intensive Periodontal Disease Treatment | Total
Number analyzed (Participants) | 17 | 34 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 25 | 40
  >=65 years | 2 | 9 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 13 | 17
  Male | 13 | 21 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 5 | 9
  Black | 5 | 19 | 24
  Hispanic | 5 | 5 | 10
  Asian | 3 | 4 | 7
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing Study Protocol
Description: The investigators will determine the number of participants who complete baseline, month 4, month 8, and month 12 study visits.
Time Frame: Baseline, Month 4, Month 8, Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Control/Delayed Treatment | Intensive Periodontal Disease Treatment
Number analyzed (Participants) | 17 | 34
Participants
  Completed Baseline Visit | 17 | 34
  Completed 4 Month Visit | 14 | 30
  Completed 8 Month Visit | 14 | 29
  Completed 12 Month Visit | 14 | 30

2. Secondary Outcome: Change in Estimated Glomerular Filtration Rate
Description: Using the creatinine-based CKD-EPI equation, the investigators will determine change in estimated glomerular filtration rate from baseline to 12 month by individual and treatment group
Time Frame: Baseline, Month 4, Month 12
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Control/Delayed Treatment | Intensive Periodontal Disease Treatment
Number analyzed (Participants) | 17 | 34
mL/min/1.73m^2
  Baseline Visit | 46.3 (10.8) | 43.4 (14.7)
  4 Month Vist | 44.7 (12.1) | 43.2 (16.6)
  12 month Visit | 45.6 (12.4) | 42.4 (18.3)

ADVERSE EVENTS:
Time Frame: Participants were asked of adverse events at their baseline, 4 month, 8 month and 12 month visits. Participants could also contact the study coordinator should any adverse events happen between visits. 3 years, 6 months
Arm/Group | Control/Delayed Treatment | Intensive Periodontal Disease Treatment
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/17 | 1/34
Other Adverse Events (participants affected / at risk) | 0/17 | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control/Delayed Treatment (N=17) | Intensive Periodontal Disease Treatment (N=34)
Minocycline Reaction (General disorders) | 0 (0) | 1 (1) — Patient reported allergic reaction, bad taste in mouth, dry socket, foul breath odor, headache, numbness, painful gums, tooth sensitivity at 8 month visit.

LIMITATIONS AND CAVEATS:
A large trial with a true control group is needed to determine the extent to which periodontal treatment may slow the trajectory of kidney function deterioration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT01802216/SAP_000.pdf
  • Study Protocol (2013-12-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT01802216/Prot_001.pdf